CLINICAL TRIAL: NCT00282113
Title: Efficacy of a Prebiotic and Probiotic Combination in Preterm Infants
Brief Title: Effects of Probiotic and Prebiotic Combinations on Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Mark A. Underwood, UC Davis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2004122333-1
Record Dates: First submitted 2006-01-23; First posted 2006-01-25 (Estimated); Results first posted 2010-01-28 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2009-12

CONDITIONS: Premature Infants; Stool Bacterial Composition; Growth
Keywords: Probiotic; Prebiotic; NEC; Premature infants; commensal flora
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ProBioPlus (Active Comparator)
  Interventions: Dietary Supplement: ProBioPlus
- Culturelle (Active Comparator)
  Interventions: Dietary Supplement: Culturelle
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: ProBioPlus — ProBioPlus is advertised as containing Lactobacillus acidophilus, Bifidobacterium longum, Bifidobacterium infantis, and Bifidobacterium bifidum plus inulin. The dose given was 5 x 10e8 twice daily.
  Arms: ProBioPlus
Dietary Supplement: Culturelle — Culturelle is advertised as containing Lactobacillus rhamnosus GG. The dose was 5 x 10e8 twice daily.
  Arms: Culturelle
Other: Placebo — A dilute preparation of pregestimil powder formulated to have a similar appearance to the probiotic products
  Arms: Placebo

SUMMARY:
The purpose of this study is to see how oral preparations containing both probiotics and prebiotics impact the growth, bacterial colonization of the intestines, and fecal short chain fatty acid content in premature infants. Our hypothesis is that short term growth will be improved, the stool will have more healthy bacteria, and the fecal short chain fatty acid content will increase in the babies who receive the probiotic/prebiotic combinations compared to control groups.

DETAILED DESCRIPTION:
Premature infants are at risk for a devastating infection of the intestines due to the immaturity of their intestines and immune system. Probiotics are bacteria with healthful qualities that are taken by mouth to improve the number of healthy bacteria in the intestines. Probiotics have been shown in several studies outside the U.S. to decrease the risk of serious intestinal infection and in one small study to improve the rate of weight gain in premature infants. Prebiotics are food supplements that stimulate the growth of healthy bacteria and suppress the growth of unhealthy bacteria. Prebiotics have been shown to improve the numbers of healthy bacteria in the stool of premature babies. Our study is designed to compare two over the counter probiotic/prebiotic combinations to each other and to a control group. Infants less than 35 weeks with a birthweight of 750-2000 gm are eligible and must be enrolled in the study within the first week of life. The babies are randomly assigned to either a control group (no probiotic/prebiotic, just a placebo), a group which receives Culturelle (Lactobacillus rhamnosus GG plus fructo-oligosaccharide, ConAgra), or a group which receives ProBioPlus (three strains of Bifidobacteria plus Lactobacillus acidophilus plus fructo-oligosaccharide, UAS Laboratories). The babies receive the study product by mouth twice daily for 28 days or until discharge (whichever comes first). Weekly measurements (weight, length, head size) and stool cultures are performed. Clinical progress is closely monitored and any episodes of infection are recorded.

ELIGIBILITY:
Inclusion Criteria:

* less than 35 weeks gestation, birth weight 750-2000 grams
* born in or transferred to University of California Davis Medical Center within first week of life
* less than eight days of age at the time of enrollment

Exclusion Criteria:

* Severe intestinal or cardiac congenital anomalies

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2004-10; Primary Completion 2006-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Sherman, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States

REFERENCES:
- [Result] Underwood MA, Salzman NH, Bennett SH, Barman M, Mills DA, Marcobal A, Tancredi DJ, Bevins CL, Sherman MP. A randomized placebo-controlled comparison of 2 prebiotic/probiotic combinations in preterm infants: impact on weight gain, intestinal microbiota, and fecal short-chain fatty acids. J Pediatr Gastroenterol Nutr. 2009 Feb;48(2):216-25. doi: 10.1097/MPG.0b013e31818de195. PMID 19179885

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Premature infants were enrolled from October 2004 to Aug 2006 at the University of California Davis Medical Center Neonatal Intensive Care Unit in Sacramento, California.
Groups:
- ProBioPlus: ProBioPlus (three bifidobacteria, Lactobacillus acidophilus, and fructo-oligosaccharide) at a dose of 5 x 10e8 organisms twice daily for five weeks
- Culturelle: Culturelle (Lactobacillus ramnosus GG plus fructo-oligosaccharide) at a dose of 5x10e8 organisms twice daily for five weeks.
- Placebo: A dilute preparation of pregestimil formula (negligible caloric content)
Period: Overall Study
Arm/Group | ProBioPlus | Culturelle | Placebo
Started | 31 | 30 | 29
Completed | 30 | 30 | 29
Not Completed | 1 | 0 | 0
Not completed — Removed at parents request | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ProBioPlus | Culturelle | Placebo | Total
Number analyzed (Participants) | 31 | 30 | 29 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31 | 30 | 29 | 90
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: weeks gestation] | 29.3 (2.6) | 29.5 (2.6) | 30.2 (2.4) | 29.7 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 10 | 31
  Male | 19 | 21 | 19 | 59
Region of Enrollment [Number; unit: participants]
  United States | 31 | 30 | 29 | 90

OUTCOME MEASURES:

1. Primary Outcome: Weight Gain
Description: Weight at five weeks minus birth weight
Time Frame: 5 weeks
Population: Infants left the study as they were discharged from the NICU, therefore many of the infants were not available for measurement at five weeks. The number reported is the number of infants remaining in the study at 5 weeks. Weight in grams is reported.
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | ProBioPlus | Culturelle | Placebo
Number analyzed (Participants) | 19 | 15 | 17
Grams | 618 (201) | 590 (186) | 682 (208)
Statistical Analysis 1: Comparison: ProBioPlus vs Culturelle vs Placebo; Test type: Superiority or Other; p > 0.5, Mixed-effects regression

2. Secondary Outcome: Stool Colonization With Bifidobacteria
Description: Using standard culture techniques, we measured how many of the first 11 infants in each arm of the study grew bifidobacteria in their feces after four weeks of treatment.
Time Frame: 4 weeks
Measure: Number; unit: Participants
Arm/Group | ProBioPlus | Culturelle | Placebo
Number analyzed (Participants) | 11 | 11 | 11
Participants | 7 | 2 | 3
Statistical Analysis 1: Comparison: ProBioPlus vs Culturelle vs Placebo; Test type: Superiority or Other; p = 0.06, Chi-squared

3. Secondary Outcome: Stool Short Chain Butyric Acid Content
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: nmoles per mg stool
Arm/Group | ProBioPlus | Culturelle | Placebo
Number analyzed (Participants) | 11 | 12 | 10
nmoles per mg stool | 5.1 (4.8) | 8.3 (5.6) | 7.7 (5.5)
Statistical Analysis 1: Comparison: ProBioPlus vs Culturelle vs Placebo; Test type: Superiority or Other; p > 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: Five weeks
Description: We found no adverse events that could be attributed to the intervention.
Arm/Group | ProBioPlus | Culturelle | Placebo
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 0/31 | 0/30 | 0/29

LIMITATIONS AND CAVEATS:
Smaller sample size than anticipated due to the number of infants enrolled who were discharged home prior to completing five weeks of treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes